CLINICAL TRIAL: NCT03901417
Title: A Randomized, Double-blind, Split-face Controlled Pilot Study to Assess the Efficacy of Combination Microneedling and Non-ablative Fractional Laser Versus Non-ablative Fractional Laser Alone for Treatment of Atrophic Acne Scars
Brief Title: Comparison of 1550nm Fractional Laser Alone Versus in Combination With Microneedling for the Treatment of Acne Scars
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Massachusetts General Hospital (Other)
Responsible Party: Principal Investigator, Mathew Avram, MD, JD, Director, Dermatologic Surgery and Laser and Cosmetic Center, Massachusetts General Hospital
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 2018P002595
Record Dates: First submitted 2019-03-26; First posted 2019-04-03 (Actual); Last update posted 2020-01-28 (Actual); Status verified 2020-01

CONDITIONS: Acne Scars

STUDY DESIGN:
Intervention Model Description: Randomized split-face clinical trial
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (2):
- Non-ablative Fractional Laser (Active Comparator): Non-ablative fractional laser (brand name Fraxel Restore) only on one half of the face.
  Interventions: Device: Fraxel Restore (Non-ablative Fractional Laser)
- Non-ablative Fractional Laser Plus Microneedling (Active Comparator): Non-ablative fractional laser (brand name Fraxel Restore) in combination with a microneedling device (SkinPen) on the other half of the face.
  Interventions: Device: Fraxel Restore (Non-ablative fractional laser) and SkinPen (Microneedling Device)

INTERVENTIONS:
Device: Fraxel Restore (Non-ablative Fractional Laser) — In the study, one side of the face will be treated with non-ablative fractional laser monthly for three months.
  Arms: Non-ablative Fractional Laser
Device: Fraxel Restore (Non-ablative fractional laser) and SkinPen (Microneedling Device) — In the study, one side of the face will be treated with a combination of non-ablative fractional laser and microneedling monthly for three months.
  Arms: Non-ablative Fractional Laser Plus Microneedling

SUMMARY:
Acne scarring is an unfortunate consequence of inflammatory acne vulgaris that often leads to significant cosmetic and psychosocial impacts. Although there have been many advances in the treatment of acne scarring, it remains one of the greatest challenges in cosmetic and laser dermatology.

There have been a multitude of studies establishing the efficacy of non-ablative fractional laser therapy for the treatment of atrophic acne scars, and it is widely regarded as one of the best available treatments. More recently, there has been a renewed interest in controlled, non-thermal dermal injury via microneedling devices in the treatment of atrophic acne scars.

Where there is a gap in the literature, however, is in the evaluation of the combination of non-ablative fractional laser resurfacing with microneedling in the treatment of atrophic acne scars.

The investigators' study will compare the safety and efficacy of using non-ablative fractional laser versus a combination of microneedling and non-ablative fractional laser for atrophic acne scars using a randomized, double-blind, split-face study.

The investigators' aim is to further elucidate the pathogenesis of acne scarring and the best approaches for treatment. In doing so, the investigators will study a combination approach to this complex problem in order to better serve future patients.

DETAILED DESCRIPTION:
Acne vulgaris is a highly prevalent dermatologic disorder that affects up to 90% percent of the population at some point in their lives to varying degrees. Acne scarring is an unfortunate complication of the inflammation that results if acne is not sufficiently treated. Classically, acne scarring has been described as either atrophic, hypertrophic, keloidal, or pigmented. Atrophic is by far the most common type of acne scarring and is subdivided into boxcar, rolling, and icepick subtypes. The presence of acne scarring has been associated with a significant decrease in patient well-being and has many psychosocial implications. Although the understanding of the pathogenesis, prevention, and treatment of acne scarring has come a long way, there are limitations to the current treatment options and the search for a cure continues.

One of the greatest advances in the treatment of acne scarring came with the advent of non-ablative fractional lasers, which work through the theory of fractional photothermolysis. Fractional photothermolysis relies on the principle of creating thousands of microthermal injury zones in the skin while allowing the surrounding intact skin to expedite wound healing. The relative sparing of the epidermis while facilitating collagen remodeling in the dermis underlies the use of non-ablative fractional laser therapy in the treatment of atrophic scars.

The erbium-doped 1,550-nm non-ablative fractional laser has been extensively studied in the treatment of atrophic acne scars with good efficacy and safety.

The concept of using needle subcision for the treatment of depressed surgical scars was first described by Orentreich et al in 1995. The first microneedling device, a drum-shaped roller was subsequently developed by Fernandes et al in the early 2000s. Several studies have validated the use of microneedling for acne scarring with a similar mechanism of creating microchannels in the dermis that allow for collagen remodeling. Furthermore, microneedling has been demonstrated to induce a specific cytokine profile including fibroblast-like growth factor, vascular endothelial growth factor, epidermal growth factor, and transforming growth factor-beta3 which are associated with favorable wound healing.

More recently, experts have advocated for the use of electric-powered microneedling devices which allow for more controlled injury at a set depth, density, and speed for the treatment of atrophic acne scars with good results.

To the investigators' knowledge, this study will be the first of its kind to compare the efficacy and safety of a combination of 1,550-nm erbium-doped fractional laser and microneedling with the SkinPenTM device to 1,550-nm erbium-doped fractional laser alone in the treatment of atrophic acne scars.

Both treatment modalities in this study are already FDA approved treatment modalities for acne scarring.

ELIGIBILITY:
Inclusion Criteria:

* All gender patients
* Age older than 18 years
* Fitzpatrick skin types I-III
* Facial acne scarring of grades III-IV
* Both sides of the face should have similar amount and severity of acne scarring

Exclusion Criteria:

* History of keloidal scarring
* Localized or active infection in the treatment region
* Immunodeficiency disorders
* Porphyria or light sensitivity
* Connective tissue disorders.
* Pregnant or nursing
* Recent isotretinoin use within the past 6 months
* Renal Disease
* Allergies to lidocaine, tetracaine, valacyclovir

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 10 (Estimated)
Dates: Start 2019-06-01 (Actual); Primary Completion 2020-06-30 (Estimated); Study Completion 2020-12-31 (Estimated)

PRIMARY OUTCOMES:
Improvement in acne scarring | 20 weeks
  Two blinded evaluators will use standardized digital photographic review to grade acne scar improvement on a quartile grading scale (1 = 1% to 25%, 2 = 26 to 50%, 3 = 51 to 75%, 4 = >76% improvement).

CONTACTS AND LOCATIONS:
Overall Officials: Mathew Avram, MD, Principal Investigator — Massachusetts General Hospital
Locations (1):
- Massachusetts General Hospital, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No